CLINICAL TRIAL: NCT04502628
Title: Hyperbaric Oxygen Therapy for the Treatment of Hemorrhagic Cystitis Post Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Hyperbaric Oxygen Therapy for Hemorrhagic Cystitis Post HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBOT for HC
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Stem Cell Transplant Complications
Keywords: allogeneic stem cell transplantation; Hemorrhagic cystitis; Hyperbaric oxygen treatment
MeSH Terms: conditions — Cystitis, Hemorrhagic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBOT group (Experimental): Patients with hemorrhagic cystitis (HC) after allo-HSCT will receive hyperbaric oxygen therapy (HBOT) on the next day of the HC diagnosis was determined. Then HBOT will be scheduled every day until symptoms of HC vanished.
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Patients with hemorrhagic cystitis (HC) after allo-HSCT will receive hyperbaric oxygen therapy (HBOT) on the next day of the HC diagnosis was determined. Then HBOT will be scheduled every day until symptoms of HC vanished. Other classic measures to treatment HC such as hydration, alkalization, and bladder irrigation will also be carried out at the same time.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative therapy for many malignant or nonmalignant hematological diseases. Hemorrhagic cystitis (HC) is one of the common and major causes of morbidity in patients undergoing allo-HSCT. Its incidence ranges from 7 to 52%, and its manifestations range from painless microscopic hematuria to severe bladder hemorrhage, leading to clot formation within the urinary tract and even renal failure. This complication results in much pain to the patient and increasing treatment cost.

Late-onset HC (two weeks after stem cell infusion) has been associated with reactivation of viruses, including cytomegalovirus, polyoma BK and JC viruses, and adenovirus types I and II. Former studies have confirmed that the bladder is also considered to be one of the immune attacked organs in acute graft-versus-host disease (aGVHD). The classic treatments for HC include hydration, alkalization, and bladder irrigation, immunosuppressant reduction, and platelet transfusion. Patients with viral infection may be treated with antiviral agents, but their efficacy is limited. When the HC was considered to be associated with aGVHD, some immunosuppressive agents such as glucocorticoids will be added in. However, too intensive immunosuppressive measures leave the patients susceptible to infection and, in turn, increases the accidence of non-relapse mortality (NRM). The mechanism underlying the development of HC remains largely unidentified, and its optimal treatment has not yet been established. It is important to explore novel, less-toxic, higher effective, and cost-effective strategies to improve HC.

The elevated levels of available oxygen and partial pressure of arterial oxygen provide the main benefits of Hyperbaric oxygen therapy (HBOT) in clinical practice that addresses these areas of inadequate or poor tissue healing. HBOT is utilized as primary or adjunctive therapy for many medical conditions in which tissue damage is triggered by hypoxic injury. The pharmacological and physiologic effects of HBOT have direct and indirect mechanisms and effects on reactive oxygen species (ROS) most beneficial to that of wound healing and antibacterial treatments. HBOT can stimulate fibroblast proliferation, angiogenesis, and wound healing. It has been shown effective in the treatment of radiation-induced HC by promoting fibroblast proliferation and capillary angiogenesis, decreasing edema, and facilitating damaged hypoxic urothelium. Based on the above clinical and pre-clinical practice, the investigators deduce that HBOT may benefit patients with HC after HSCT. In the investigators' limited early-onset investigation, the investigators found HBO was largely successful in 20 patients suffering HC post-allo-HSCT, showed a quick resolution or improvement of HC. The investigators also observed more rapid responses in patients who started HBOT earlier after the diagnosis of HC. The investigators confirmed that HBOT was effective and well-tolerated in the patients, regardless of the infective- or non-infective- caused HC. Therefore, the investigators design this prospective, randomized, and single-arm clinical trial to establish the definitive efficacy and safety of HBOT in patients with HC after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing allogeneic stem cell transplantation
* Patients develop late-onset hemorrhagic cystitis (HC)
* The count of neutrophilia cells over 0.5 * 10^9/L, hemoglobin over 60 g/L, platelet over 30 *10^9/L
* SGOT/SGPT no more than 2 times of UNL
* Serum creatinine no more than 1.5 times of UNL
* Signed informed consent

Exclusion Criteria:

* Early-onset HC post-allo-HSCT
* Unsuitable to the study due to severe complication such as uncontrolled severe infection
* Claustrophobia
* Ear diseases such as otitis media
* Eye diseases such as glaucoma
* Epilepsy history
* Important organ dysfunction
* Coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate of HBOT | Six months post-allo-HSCT
  Response rate of HBOT was determined on the basis of HC symptom disppearance and the normal urine routine test result
Incidence and severity of treatment-related adverse events | 3 years
  Number of participants with treatment-related adverse events and the the severity of these events.

SECONDARY OUTCOMES:
Exploratory biomarker analysis | 3 years
  Exploratory biomarker to predict treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue C, Chen H, Zhao Y, Yuan D, Fang X, Ding M, Qu H, Wang X, Ge X, Lu K, Jiang Y. Preventive hyperbaric oxygen therapy improves acute graft-versus-host disease by activating the Nrf2/HO-1 pathway. Front Immunol. 2025 Feb 27;16:1529176. doi: 10.3389/fimmu.2025.1529176. eCollection 2025. PMID 40083556